CLINICAL TRIAL: NCT07264543
Title: Evaluation of Early Methylene Blue in the Microhemodynamics of Septic Shock Patients: a Feasibility Randomized Controlled Trial
Brief Title: Early Methylene Blue in the Microhemodynamics of Septic Shock Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro de Estudos e Pesquisa em Emergencias Medicas e Terapia Intensiva (Other)
Collaborators: Irmandade da Santa Casa de Misericordia de Curitiba (Other)
Responsible Party: Principal Investigator, Bruna Cassia Dal Vesco, Clinical Research Fellow, Centro de Estudos e Pesquisa em Emergencias Medicas e Terapia Intensiva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1331-7627; Approval number 7.955.174 (Other: Pontifícia Universidade Católica do Paraná - Research and Ethics Committee); CAAE 93099325.5.0000.0020 (Other: Pontifícia Universidade Católica do Paraná - Research and Ethics Committee)
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Septic Shock; Hypoperfusion
Keywords: Septic Shock; Methylene Blue; Microcirculation; Capillary Refill Time
MeSH Terms: conditions — Shock, Septic | interventions — Methylene Blue; Phenothiazines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the high probability of the intervention group present blue coloured skin and secretions caused by MB infusion, the study is classified as open-label for patients, assisting staff and investigators. Blinding remains for the team that will perform the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene blue group (Experimental): The intervention group will receive methylene blue plus standard treatment for septic shock, according to the international guidelines.
  Interventions: Drug: Methylene blue infusion
- Control group (No Intervention): The control group will receive the standard treatment according to international guidelines for the management of sepsis and septic shock.

INTERVENTIONS:
Drug: Methylene blue infusion — Methylene blue at a dose of 100mg (diluted in 100ml of 5% dextrose solution) in continuous infusion for 06 hours per day, for 03 days, plus standard treatment according to international guidelines for the management of sepsis and septic shock. The 03 consecutive MB infusions, each lasting 06 hours, will be performed every 24 hours, starting from randomization: the first infusion at T0, the second at T24, and the third at T48, considering T0 the moment after the patient randomization into the study.
  The interruption of the protocol will be recommended if vasopressors are completely discontinued during the three days of methylene blue infusion. The attending physician may discontinue methylene blue treatment if judges necessary. Similarly, interruption may occur if the family or patient request.
  Other Names: Methylene blue; Phenothiazines
  Arms: Methylene blue group

SUMMARY:
The aim of the study is to evaluate the viability and feasibility of its protocol in order to conduct a larger clinical trial to assess whether methylene blue can improve patient-centered clinical outcomes such as mortality or length of hospital stay in septic shock patients.

DETAILED DESCRIPTION:
One of the primary causes of high mortality in patients with septic shock is microcirculatory dysfunction related to vasodilation caused by excessive oxide nitric production. It has been shown that methylene blue, an old and safe drug that can reduce vasodilation by blocking nitric oxide pathways, is a vasopressor-sparing treatment in sepsis. Nevertheless, there is no evidence that methylene blue improves patient-centered clinical outcomes such as mortality. Understanding how early methylene blue affects the microhemodynamics of septic shock patients may lead to relevant clinical results that can improve their prognosis. So, the objective of the study is to evaluate the viability and feasibility of the study protocol for a larger clinical trial, assessing the effectiveness of early methylene blue in the microhemodynamics of septic shock patients, mainly through the capillary refill time measurement. For this purpose, a pilot study of an open-label, randomized, controlled and single-center clinical trial will be conducted, with two treatment arms: the intervention group (methylene blue plus standard treatment) and the control group (standard treatment). Fifty adult patients with septic shock within the first six hours of diagnosis will be included in this study. They will be randomized to either receive a methylene blue infusion or not. The randomization will be conducted using RedCap with a 1:1 ratio and variable block sizes. The primary outcome will be to assess the feasibility, which is defined as completing the study recruitment within the 12-month timeline and achieving protocol adherence of 90% or higher. Comparisons between groups for serially measured micro and macrohemodynamics parameters will be the secondary outcomes. Additionally, the incidence of adverse events related to methylene blue will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with septic shock according to SEPSIS-3 definition, within less than 6 hours of the diagnosis.

Exclusion Criteria:

* Pregnant or breastfeeding patients;
* Patients with any withdrawal or withholding life-sustaining intervention;
* Cardiac surgery patients in the immediate postoperative period;
* Personal or familiar history of glucose-6-phosphate dehydrogenase (G6PD) deficiency;
* Allergy to methylene blue, phenothiazines, or food dyes;
* Recent administration of linezolid (less than 14 days ago);
* Recent intake of serotonergic psychiatric medications (less than 2 weeks ago - with the exception of fluoxetine, which must be less than 5 weeks ago),
* Recent intake (less than 2 weeks ago) of monoamine oxidase inhibitors (MAOIs), such as rasagiline and selegiline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of the study protocol. | 28 days after randomization.
  The primary outcome of the study is to evaluate feasibility, defined as completing the study protocol according to the planned timeline and with 90% or more protocol adherence. Protocol adherence will be defined as the use of the allocated therapy in the intervention group for 6 hours for 3 days (or interruption of methylene blue if the patient does not require a vasoactive drug anymore). Justified interruptions will not be considered violations.

SECONDARY OUTCOMES:
Capillary refill time | 72 hours after randomization.
  Serial capillary refill time from randomization up to 72 hours later.
Serum lactate level | 72 hours after randomization.
  Serial measurements of serum lactate level during the 72 hours after randomization.
Arteriovenous carbon dioxide difference (gapCO2) | 72h after randomization.
  Serial measurements of arteriovenous carbon dioxide difference (gapCO2) during 72h after randomization.
Central venous oxygen saturation (SvO2) | 72h after randomization.
  Serial measurements of central venous oxygen saturation (SvO2) during 72h after randomization.
Serial measurements of heart rate | 72 hours after randomization.
  Serial measurements of heart rate from randomization up to 72 hours later.
Serial measurements of mean arterial pressure | 72 hours after randomization.
  Serial measurements of mean arterial pressure from randomization up to 72 hours later.
Serial measurements of pulse pressure | 72 hours after randomization.
  Serial measurements of pulse pressure from randomization up to 72 hours later.
Serial measurements of systolic arterial pressure | 72 hours after randomization.
  Serial measurements of systolic arterial pressure from randomization up to 72 hours later.
Serial measurements of dyastolic arterial pressure | 72 hours after randomization.
  Serial measurements of dyastolic arterial pressure from randomization up to 72 hours later.
Methylene blue-related adverse events | 28 days after randomization.
  Incidence of adverse events during the three days of administration of methylene blue and up to 28 days after.

OTHER OUTCOMES:
Variations in the Sequential Organ Failure Assessment-2 Score (SOFA-2) | From enrollment to 72 hours later.
  Daily SOFA-2 score pontuatin from enrollment to 72 hours later. The SOFA score ranges from 0 to 24, being 24 the worst pontuation, indicating multiple organ dysfunction.
Time to vasopressor discontinuation | 28 days after randomization.
  Time to complete vasopressor discontinuation from the enrollment up to 28 days.
Vasopressor dose (norepinephrine and vasopressin) | 72 hours after randomization.
  Vasopressor dose (norepinephrine and vasopressin) before and after the start of MB infusion, measuring before and after the methylene blue on the first, second, and third days of infusion.
Time to weaning from mechanical ventilation | 28 days after randomization.
  Total number of days to wean from mechanical ventilation during the 28 days after randomization.
Need for renal replacement therapy (RRT) | 28 days after randomization.
  Total number of days of renal replacement therapy (RRT) during 28 days after randomization.
Intensive care unit length of stay | 28 days after randomization.
  Total number of days until intensive care unit discharge.
28-day mortality | 28 days after randomization.
  All-cause mortality at day 28 after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Réa-Neto, Study Chair — CEPETI - Centro de Estudos e Pesquisa em Emergências Médicas e Terapia Intensiva
Locations (1):
- Irmandade da Santa Casa de Misericórdia de Curitiba, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No